CLINICAL TRIAL: NCT05742321
Title: Analysis of the Genotype/Phenotype Relationship in the Fuchs' Corneal Endothelial Dystrophy in France. The French Fuchs' Follow-up Study (Phase 2), F3S2
Brief Title: Analysis of the Genotype/Phenotype Relationship in the Fuchs' Corneal Endothelial Dystrophy in France
Acronym: F3S2
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Kyoto University, Graduate School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 22CH354; 2022-A01217-36 (Other: ANSM)
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Corneal Dystrophies
Keywords: Corneal Dystrophies; Corneal Endothelial Dystrophy; Fuchs' Corneal Endothelial Dystrophy, FECD
MeSH Terms: conditions — Corneal Dystrophies, Hereditary; Corneal Dystrophy, Posterior Polymorphous, 1; Fuchs' Endothelial Dystrophy | interventions — Genotype; Shadowing Technique, Histology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample will be performed (genetic analyses)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with FECD: Patients with Fuchs Endothelial Corneal Dystrophy (FECD). They will have a collection of data and a blood sample
  Interventions: Genetic: Genotyping; Diagnostic Test: Histology; Other: Collection of data

INTERVENTIONS:
Genetic: Genotyping — Genotyping will measure the triple nucleotide repeat in the TCF4 gene and search for other known mutations in other genes Blood sample will be performed (genetic analyses).
Diagnostic Test: Histology — Histology will be performed on flat mounted Descemet membrane obtained after Descemetorhexis
Other: Collection of data — Collection of data of examination for diagnosis of the Fuchs Endothelial Corneal Dystrophy (FECD) including slit lamp results will be performed.

SUMMARY:
The pathophysiology of the most common corneal endothelial dystrophies (Fuchs' Corneal Endothelial Dystrophy, FECD) is beginning to be dismembered. There is a significant heterogeneity in the clinical forms and the investigators have just highlighted a great diversity of histological forms that seem to define distinct groups.

DETAILED DESCRIPTION:
The most frequent genetic abnormalities have been published since 10 years and can now be easily searched. This study is going to analyze the relationships between clinical, histological and genetic forms in a large population to better understand how histological abnormalities are formed.

ELIGIBILITY:
Inclusion Criteria:

* affiliated with or entitled to a social security scheme
* Consent form to participate in the study signed
* with an FECD certified by slit lamp examination
* requiring an endothelial keratoplasty

Exclusion Criteria:

- Patients under guardianship or curators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with FECD as evidenced by slit lamp examination and scheduled for endothelial transplantation within one quarter of inclusion;
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of CTG triplet repetitions in the intron of the Transcription Factor 4 (TCF4) gene | At inclusion
  Polymerase Chain Reaction (PCR) will be performed from DNA (blood sample)

SECONDARY OUTCOMES:
Refraction with the auto-refractor tonometry | At inclusion
  Analysis refraction with the auto-refractor tonometry non-contact air.
ETDRS scale (international standardized Early Treatment Diabetic Retinopathy Study scale) | At inclusion
  ETDRS (Early Treatment Diabetic Retinopathy Study) scale will be allowed to measure visual acuity uses an eye chart with 5 letters per line. The scores range from 0 (no letters read correctly) to 100 (all letters read correctly).
Corneal thickness in Optical Coherence Tomography (OCT) | At inclusion
  Corneal thickness measured by OCT in micrometers
Diameter of the dilated pupil (mm) | At inclusion
  Measured by contact or non-contact biometry
Thickness of the lens (mm) | At inclusion
  Measured by contact or non-contact biometry
Depth of the anterior chamber (mm) | At inclusion
  Measured by contact or non-contact biometry
Endothelial cell density measurement (cells/mm2) | Immediately after surgery of corneal transplantation"
  Endothelial cell density (cells/mm2) in the center and in the 4 standardized cardinal positions high low nasal temporal.
Crystalline analysis | Immediately after surgery of corneal transplantation"
  Crystalline : clear lens, cataract, intraocular implant, aphakic
Family cases of Fuchs' Corneal Endothelial Dystrophy | At inclusion
  Family cases: absent/probable/advanced
Frequency of the mutation rs613872 in the intron of the Transcription Factor 4 (TCF4) gene. | At inclusion
  PCR reactions will be performed from DNA (blood sample)

CONTACTS AND LOCATIONS:
Overall Officials: GILLES THURET, MD-PhD, Principal Investigator — CHU DE SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No